CLINICAL TRIAL: NCT03564886
Title: Safety and Efficacy of Hyperosmolar Saline Irrigation Fluid in Arthroscopic Knee Surgery
Brief Title: Hyperosmolar Saline Irrigation Fluid in Arthroscopic Knee Surgery
Acronym: Salty Knee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, James Stannard, Hansjörg Wyss Distinguished Chair in Orthopaedic Surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011296
Record Dates: First submitted 2018-06-08; First posted 2018-06-21 (Actual); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Arthroscopic Knee Surgery
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperosmolar Saline (Experimental): The hyperosmolar solution will be created by adding 120cc of 23.4% NS solution to a 3L bag of LR.
  Interventions: Drug: Hyperosmolar Saline
- Normal Saline (Placebo Comparator): Lactate Ringer's (LR, 273mOsm/L) is commonly used at our facility as our isotonic standard irrigation solution and will serve as the control to be evaluated against a hyperosmolar (1.9%, 600mOsm) solution.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Hyperosmolar Saline — The hyperosmolar solution will be created by adding 120cc of 23.4% NS solution to a 3L bag of LR.
  Arms: Hyperosmolar Saline
Drug: Normal saline — Lactate Ringer's (LR, 273mOsm/L)
  Arms: Normal Saline

SUMMARY:
An isotonic solution, such as saline (0.9%, 300mOsm/L) or lactated ringer's (273 mOsm/L), is commonly used and safely proven for joint irrigation during arthroscopy. Arthroscopic fluid is usually pressurized to enable visualization through dilation of the joint or bursa and prevent bleeding from the microvasculature. It has been recommended that this pressure be maintained at 49mmHg or less below the systolic blood pressure to preserve the clarity of view. The combination of large amounts of pressurized irrigation solution and lengthy arthroscopic procedures may cause substantial tissue fluid retention. Thus, extravasation of irrigation fluid into the periarticular tissues is inevitable and may create technical difficulties as well as patient morbidity and complications. Previous investigators have reported complications including tracheal obstruction, post-operative airway edema and compromise leading to prolonged intubation, excess weight gain, neurologic injuries, skin necrosis, and fluid overload associated with excessive fluid extravasation and tissue retention. Furthermore, it has been shown that fluid accumulated during the operation is slowly released back into the systemic circulation. Although there is not a rapid change in circulating volume, there may be implications for elderly patients and those with multiple comorbidities during prolonged arthroscopic surgery. Therefore the investigators seek to determine if a hyperosmolar solution, similar to what is used in head trauma patients, can reduce the degree of fluid extravasation in knee arthroscopy. The investigators also seek to determine if a hyperosmolar solution has any effect on post-operative knee pain compared to the standard isotonic solution. The third objective is to determine if a hyperosmolar solution has any effect on post-operative pain medicine consumption compared to the standard isotonic solution.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age or greater) undergoing arthroscopic knee surgery who are willing and able to consent.

Exclusion Criteria:

* Current pregnancy or breastfeeding
* Unable to give consent
* Prisoner
* Mentally Disabled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James P Stannard, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Health System, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hyperosmolar Saline | Normal Saline
Started | 24 | 24
Completed | 23 | 23
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyperosmolar Saline | Normal Saline | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (12.5) | 44.0 (13.8) | 42.1 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 8 | 11 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (7.1) | 31.7 (6.9) | 31.0 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Fluid Extravasation
Description: To determine if a hyperosmolar solution, similar to what is used in head trauma patients, can change the degree of fluid extravasation in knee arthroscopy.
Time Frame: Immediately Postoperatively
Population: Change in Knee Girth (cm)= Postoperative knee girth- preoperative knee girth
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Hyperosmolar Saline | Normal Saline
Number analyzed (Participants) | 23 | 23
centimeters | 1.8 (1.1) | 1.2 (1.1)

2. Secondary Outcome: Postoperative Pain
Description: To determine if a hyperosmolar solution has any effect on post-operative knee pain (Visual Analogue Scale; 0-10; 0= no pain; 10= worst pain imaginable) compared to the standard isotonic solution.
Time Frame: Post-operative Days 1, 2 and 3
Population: Visual Analogue Score (0-10) for the first three postoperative days.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hyperosmolar Saline | Normal Saline
Number analyzed (Participants) | 23 | 23
units on a scale
  VAS Pain PostOp Day 1 | 4.9 (2.0) | 4.8 (2.0)
  VAS Pain PostOp Day 2 | 3.8 (1.7) | 4.8 (2.5)
  VAS Pain PostOp Day 3 | 3.6 (1.9) | 3.8 (1.7)

3. Secondary Outcome: Opioid Consumption
Description: To determine if a hyperosmolar solution has any effect on post-operative pain medicine consumption compared to the standard isotonic solution.
Time Frame: Postoperative Days 1, 2 and 3.
Population: Pain medication consumption on postoperative days 1, 2, and 3 as measured in morphine equivalent units
Measure: Mean (Standard Deviation); unit: morphine equivalent units
Arm/Group | Hyperosmolar Saline | Normal Saline
Number analyzed (Participants) | 23 | 23
morphine equivalent units
  Medication PostOp Day 1 | 17.0 (14.9) | 23.6 (18.3)
  Medication PostOp Day 2 | 15.0 (19.7) | 19.5 (18.4)
  Medication PostOp Day 3 | 4.0 (7.6) | 15.5 (17.4)

ADVERSE EVENTS:
Time Frame: 30 Days
Description: A member of the research team was responsible for documenting any perioperative adverse events that occurred prior to discharge. A retrospective review of the electronic medical records was performed to identify any adverse events that occurred within the first 30 days following surgery.
Arm/Group | Hyperosmolar Saline | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 1/23 | 0/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyperosmolar Saline (N=23) | Normal Saline (N=23)
Deep Vein Thrombosis (DVT) (Vascular disorders) | 1 (1) | 0 (0) — Post-operative DVT

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT03564886/Prot_001.pdf